CLINICAL TRIAL: NCT00700258
Title: STAR-TOR- REGISTRY FOR THE EVALUATION OF THE SAFETY, TOLERABILITY AND EFFICACY OF TEMSIROLIMUS (TORISEL), SUNITINIB (SUTENT) AND AXITINIB (INLYTA) FOR THE TREATMENT OF SUBJECTS WITH ADVANCED RENAL CELL CARCINOMA (MRCC), MANTLE CELL LYMPHOMA (MCL) AND GASTRO-INTESTINAL STROMA TUMOR (GIST).
Brief Title: Registry For Temsirolimus, Sunitinib, And Axitinib Treated Patients With Metastatic Renal Cell Carcinoma (mRCC), Mantle Cell Lymphoma (MCL), And Gastro-Intestinal Stroma Tumor (GIST) [STAR-TOR]
Acronym: STAR-TOR
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3066K1-4407; B1771009 (Other: Alias Study Number)
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Renal Cell, Advanced; Lymphoma, Mantle-Cell; Gastrointestinal Stroma Tumors
MeSH Terms: conditions — Carcinoma; Lymphoma, Mantle-Cell | interventions — temsirolimus; Sunitinib; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Patients treated with Temsirolimus for metastatic renal cell carcinoma (mRCC) under usual care settings.
  Interventions: Drug: Temsirolimus
- 2: Patients treated with Temsirolimus for mantle cell lymphoma (MCL) under usual care setting
  Interventions: Drug: Temsirolimus
- 3: Patients treated with Sunitinib for metastatic renal cell carcinoma (mRCC) under usual care setting
  Interventions: Drug: Sunitinib
- 4: Patients treated with Sunitinib for gastro-intestinal stroma tumor (GIST) under usual care setting
  Interventions: Drug: Sunitinib
- 5: Patients treated with Axitinib after treatment with Sunitinib or Cytokine for metastatic renal cell carcinoma (mRCC)
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Temsirolimus — Non-interventional study. Treatment decision already made before inclusion into the registry.
  Groups: 1
Drug: Temsirolimus — Non-interventional study. Treatment decision already made before inclusion into the registry.
  Groups: 2
Drug: Sunitinib — Non-interventional study. Treatment decision already made before inclusion into the registry.
  Groups: 3
Drug: Sunitinib — Non-interventional study. Treatment decision already made before inclusion into the registry.
  Groups: 4
Drug: Axitinib — Non-interventional study. Treatment decision already made before inclusion into the registry.
  Groups: 5

SUMMARY:
The purpose of this registry is to obtain a general view as regards efficacy, tolerability and safety issues of the Torisel®, Sutent®, and/or Inlyta® therapies in patients with advanced renal cell carcinoma, recurrent / refractory mantle cell lymphoma (MCL) and gastro-intestinal stroma tumors (GIST) under the conditions of routine use

DETAILED DESCRIPTION:
Treatment of the metastatic renal cell carcinoma (mRCC) has experienced fundamental changes within a very short period of time. In the past few years, introduction of various new substances for the treatment of mRCC has therefore resulted in new scientific research questions. Temsirolimus and sunitinib are current standard therapies in the first-line treatment of mRCC. Inlyta® is a new substance that was developed for the treatment of mRCC after failure of sunitinib or cytokines.

Since August 2009, Torisel® is available as another treatment option for patients with mantle cell lymphoma (MCL). In addition, Sutent® is used for patients with non-resectable / metastatic gastro-intestinal stroma tumors (GIST) after failure or intolerability of imatinib.

The routine use of drugs in the usual clinical setting faces additional challenges that generally cannot be completely reflected by clinical trials. Therefore, the purpose of this registry is to obtain a general view as regards efficacy, tolerability and safety issues of the Torisel®, Sutent®, and/or Inlyta® therapies in patients with advanced renal cell carcinoma, recurrent / refractory mantle cell lymphoma (MCL) and gastro-intestinal stroma tumors (GIST) under the conditions of routine use.

Therefore, the following information is of particular interest in the course of the investigation:

* Efficacy (best response, overall survival, progression-free survival)
* Tolerability of the therapy (assessed by the physician)
* Safety profile (overall incidence of adverse events as well as side-effect rate) of subjects with mRCC, rMCL, and GIST under treatment with Torisel®, Sutent®, and/or Inlyta®
* Profile, comorbidities, and characteristics of subjects treated with Torisel® Sutent®, and/or Inlyta®
* The sequence of using the systemic therapies for RCC, MCL, and GIST
* Patient survey on the quality of life of mRCC patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven tumor of RCC, MCL or GIST by histology.
* Informed consent signed by patient.

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumor patients with renal cell carcinoma (RCC), mantle cell lymphoma (MCL) or gastro-intestinal stroma tumor (GIST)
  Gastro-Intestinal Stroma Tumor
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Actual)
Dates: Start 2008-02-13 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (77):
- Germany (77):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Dr. med. Harald Held, Neumünster, Schleswig-Holstein
  - Dr. med. Hans Wilhelm Duebbers, Ahaus
  - Dr. Ludwig Fischer von Weikersthal, Amberg
  - Group Practice Doctors Klausmann, Aschaffenburg
  - Studienzentrum Drs. Klausmann / Dr. Welslau, Haematologie-Onkologie-Diabetologie, Aschaffenburg
  - Office of Detlef Muller, Bautzen
  - Medilei GmbH, Bayreuth
  - Universitaetsklinikum Charite Campus, Berlin
  - Carsten Lange, Bernburg
  - Office of Axel Belusa, Chemnitz
  - Office of Ulrich Kube, Chemnitz
  - Dr. Jens-Uwe Krieger, Chemnitz
  - Zeisigwaldklinikum Bethanien Chemnitz, Chemnitz
  - Steinmetz, Cologne
  - Klinisches Studienzentrum Urlogie, Cologne
  - Leonhard Stark, Deggendorf
  - Prof. Dr. med. Udo Rebmann, Dessau
  - doctor's office Dr. Göhler, Dresden
  - Dr.med Johannes Mohm, Dresden
  - Dr. med. Ralf Eckert, Eisleben Lutherstadt
  - Specialist Urology, Erfurt
  - Goebell, Erlangen
  - Prof. Dr. med. Lothar Bergmann, Frankfurt am Main
  - Dr. med. Gunter Derigs, Frankfurt am Main
  - Hoffkes, Fulda
  - Dr. med. Arne Strauss, Göttingen
  - PD Dr. Uwe Zimmermann, Greifswald
  - Internistische Gemeinschaftspraxis, Güstrow
  - Dr. med. Michael Rink, Hamburg
  - Office of Oleg Rubanov, Hamelin
  - Dr. med. Hanns-Detlev Harich, Hof
  - Universitaetsklinikum des Saarlandes, Klinik fuer Urologie und Kinderurologie, Homburg/Saar
  - Dr. med. Susan Foller, Jena
  - Office of Richard Hansen, Kaiserslautern
  - Dr. med. Martina Stauch, Kronach
  - Dr. med. Ursula Vehling-Kaiser, Landshut
  - Dr. Andreas Kohler, Langen
  - Dietel, Leipzig
  - Andreas Schwarzer, Leipzig
  - Resident Doctor, Leipzig
  - DRK Krankenhaus Luckenwalde, Luckenwalde
  - Dr.med. Matthias Schulze, Markkleeberg
  - Institut of Healthcare Research, Mayen
  - OnkoLog GbR, Moers
  - Stauferklinikum Schwaebisch Gmuend, Mutlangen
  - Dr. med. Jan Klaus Schroder, Mülheim
  - Dr.med. Wolfgang Abenhardt, München
  - Boegemann, Münster
  - Dr. med. Thomas Gehring, Neckarsulm
  - Dres. Derouet Poenicke Becker, Neunkirchen
  - Physician for Internal Medicine, Neuwied
  - Dr. med. David Kunst, Nienburg
  - Dr.med. Christian Linder, Nordhausen
  - Dr. med. Joachim Zimber, Nuremberg
  - Ralf-Bodo Kühn, Oldenburg
  - Prof. Dr. med. Ruhnke, Osnabrück
  - Dr. med. Torsten Geyer, Ostfildern
  - Dr. med. Ino Kietz, Parchim
  - Praxis, Plauen
  - Oncologianova GmbH, Recklinghausen
  - Andreas Hübner, Rostock
  - Facharzt für Internistische Onkologie, Hämatologie und Hämostaseologie, Saalfeld
  - Diakonie-Klinikum gGmbH, Schwäbisch Hall
  - Dr. med. Thomas Geer, Schwäbisch Hall
  - MVZ Kloster Paradiese GbR, Soest
  - Office of Judith Franz-Werner, Speyer
  - Dr. Matthias Groschek, Stolberg
  - Dr. med. Heinz Kirchen, Trier
  - Klinik für Urologie, Eberhard-Karls-Universitaet Tuebingen,, Tübingen
  - Klotz, Weiden
  - Dr.med. Jan Janssen, Westerstede
  - ZAS - Zentrum fuer angewandte Studien, Wilhelmshaven
  - Jochen Gleissner, Wuppertal
  - Universitaetsklinik Wuerzburg, Medizinische Poliklinik, Würzburg
  - Mathias Schulze, Zittau
  - Scheffler, Zwickau

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Uhlig A, Bergmann L, Bogemann M, Fischer T, Goebell PJ, Leitsmann M, Reichert M, Rink M, Schlack K, Trojan L, Uhlig J, Woike M, Strauss A. Sunitinib for Metastatic Renal Cell Carcinoma: Real-World Data from the STAR-TOR Registry and Detailed Literature Review. Urol Int. 2024;108(3):198-210. doi: 10.1159/000536563. Epub 2024 Feb 2. PMID 38310863
- [Derived] Strauss A, Schmid M, Rink M, Moran M, Bernhardt S, Hubbe M, Bergmann L, Schlack K, Boegemann M. Real-world outcomes in patients with metastatic renal cell carcinoma according to risk factors: the STAR-TOR registry. Future Oncol. 2021 Jun;17(18):2325-2338. doi: 10.2217/fon-2020-1020. Epub 2021 Mar 16. PMID 33724867
- [Derived] Boegemann M, Schlack K, Rink M, Bernhardt S, Moran M, Hubbe M, Bergmann L, Schmid M, Strauss A. Effect of comorbidities/comedications on sunitinib outcomes for metastatic renal cell carcinoma: the STAR-TOR registry. Future Oncol. 2020 Dec;16(35):2939-2948. doi: 10.2217/fon-2020-0548. Epub 2020 Oct 6. PMID 33021843
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-4407&StudyName=Registry%20For%20Temsirolimus%2C%20Sunitinib%2C%20And%20Axitinib%20Treated%20Patients%20With%20Metastatic%20Renal%20Cell%20Carcinoma%20%28mRCC%29%2C%20Mantle%20Cell%20Lymp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from eligible participants diagnosed with metastatic renal cell carcinoma (mRCC), relapsed or refractory mantle cell lymphoma (MCL) or gastrointestinal stromal tumors (GIST) and who were treated with temsirolimus, sunitinib and/or axitinib, as per routine clinical practice from January 2008 to December 2021 were observed in this prospective, non-interventional, STAR-TOR registry study.
Groups:
- Participants With mRCC, MCL or GIST: Participants diagnosed with mRCC, MCL or GIST who received temsirolimus, sunitinib and/or axitinib from January 2008 to December 2021 (approximately 14 years), as per routine clinical practice. Due to the non-interventional nature of the registry, no specific requirements were applied regarding the management of treatment. Dosing and duration of treatment was decided by the physician according to individual treatment requirements of the participant. Summary of product characteristics was considered: the daily dose of temsirolimus for mRCC participants was either 25 milligrams (mg) or 50 mg once per week and for MCL participants was 175 mg for first 3 weeks and later reduced to 75 mg. The daily dose for sunitinib should not exceed 75 mg or drop below 25 mg; the recommended starting dose of axitinib was 5 mg twice daily. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with temsirolimus, sunitinib or axitinib was discontinued or documentation was stopped for any reason.
Period: Overall Study
Arm/Group | Participants With mRCC, MCL or GIST
Started | 1520
Participants With mRCC | 1435
Participants With MCL | 59
Participants With GIST | 26
Participants With mRCC Who Received Temsirolimus | 605
Participants With mRCC Who Received Sunitinib | 702
Participants With mRCC Who Received Axitinib | 237
Participants With MCL Who Received Temsirolimus | 59
Participants With GIST Who Received Sunitinib | 26
Completed | 289
Not Completed | 1231
Not completed — Premature discontinuation of documentation | 136
Not completed — Type of study end not documented | 1
Not completed — Lost to Follow-up | 81
Not completed — Premature discontinuation of therapy | 1013

BASELINE CHARACTERISTICS:
Population: Safety analysis set comprised of all prospectively documented participants with a histologically proven diagnosis of either mRCC, MCL or GIST and at least 1 documented administration of temsirolimus, sunitinib or axitinib or any non-Pfizer treatment. Participants mentioned here are not exclusive to one treatment, one participant could have received more than one treatment.
Groups:
- Participants With mRCC, MCL or GIST: Participants diagnosed with mRCC who received only temsirolimus from January 2008 to December 2021, as per routine clinical practice were observed during this prospective registry study. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with temsirolimus was discontinued or documentation was stopped for any reason.
Arm/Group | Participants With mRCC, MCL or GIST
Number analyzed (Participants) | 1520
Age, Customized [Count of Participants; unit: Participants] — Population: Participants mentioned here are not exclusive to one treatment, one participant could have received more than one treatment.
  Participants
    mRCC - Temsirolimus: number analyzed (Participants) | 605
    mRCC - Temsirolimus: Less than (<) 40 years | 2
    mRCC - Temsirolimus: 40 - <50 years | 34
    mRCC - Temsirolimus: 50 - <60 years | 106
    mRCC - Temsirolimus: 60 - <70 years | 188
    mRCC - Temsirolimus: 70 - <80 years | 238
    mRCC - Temsirolimus: 80 - <90 years | 36
    mRCC - Temsirolimus: 90 - <100 years | 0
    mRCC - Temsirolimus: Missing | 1
    mRCC - Sunitinib: number analyzed (Participants) | 702
    mRCC - Sunitinib: Less than (<) 40 years | 5
    mRCC - Sunitinib: 40 - <50 years | 29
    mRCC - Sunitinib: 50 - <60 years | 128
    mRCC - Sunitinib: 60 - <70 years | 222
    mRCC - Sunitinib: 70 - <80 years | 252
    mRCC - Sunitinib: 80 - <90 years | 66
    mRCC - Sunitinib: 90 - <100 years | 0
    mRCC - Sunitinib: Missing | 0
    mRCC - Axitinib: number analyzed (Participants) | 237
    mRCC - Axitinib: Less than (<) 40 years | 3
    mRCC - Axitinib: 40 - <50 years | 5
    mRCC - Axitinib: 50 - <60 years | 47
    mRCC - Axitinib: 60 - <70 years | 67
    mRCC - Axitinib: 70 - <80 years | 92
    mRCC - Axitinib: 80 - <90 years | 23
    mRCC - Axitinib: 90 - <100 years | 0
    mRCC - Axitinib: Missing | 0
    MCL - Temsirolimus: number analyzed (Participants) | 59
    MCL - Temsirolimus: Less than (<) 40 years | 0
    MCL - Temsirolimus: 40 - <50 years | 0
    MCL - Temsirolimus: 50 - <60 years | 3
    MCL - Temsirolimus: 60 - <70 years | 11
    MCL - Temsirolimus: 70 - <80 years | 33
    MCL - Temsirolimus: 80 - <90 years | 11
    MCL - Temsirolimus: 90 - <100 years | 1
    MCL - Temsirolimus: Missing | 0
    GIST - Sunitinib: number analyzed (Participants) | 26
    GIST - Sunitinib: Less than (<) 40 years | 1
    GIST - Sunitinib: 40 - <50 years | 1
    GIST - Sunitinib: 50 - <60 years | 3
    GIST - Sunitinib: 60 - <70 years | 7
    GIST - Sunitinib: 70 - <80 years | 12
    GIST - Sunitinib: 80 - <90 years | 2
    GIST - Sunitinib: 90 - <100 years | 0
    GIST - Sunitinib: Missing | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Participants mentioned here are not exclusive to one treatment, one participant could have received more than one treatment.
  Participants
    mRCC - Temsirolimus: number analyzed (Participants) | 605
    mRCC - Temsirolimus: Male | 410
    mRCC - Temsirolimus: Female | 191
    mRCC - Temsirolimus: Missing | 4
    mRCC - Sunitinib: number analyzed (Participants) | 702
    mRCC - Sunitinib: Male | 510
    mRCC - Sunitinib: Female | 187
    mRCC - Sunitinib: Missing | 5
    mRCC - Axitinib: number analyzed (Participants) | 237
    mRCC - Axitinib: Male | 163
    mRCC - Axitinib: Female | 71
    mRCC - Axitinib: Missing | 3
    MCL - Temsirolimus: number analyzed (Participants) | 59
    MCL - Temsirolimus: Male | 41
    MCL - Temsirolimus: Female | 18
    MCL - Temsirolimus: Missing | 0
    GIST - Sunitinib: number analyzed (Participants) | 26
    GIST - Sunitinib: Male | 17
    GIST - Sunitinib: Female | 8
    GIST - Sunitinib: Missing | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from initiation of treatment to death from any cause. In case a death was documented, but date of death was unknown, the date of death was substituted with the latest available date for the participant (last visit, last contact date, date of assessment). If no death was documented, participant was censored with the latest available contact date or assessment date within study. If these rules led to a missing duration or a negative duration, duration was set to maximum of (PFS,"1 day"). Progression free survival (PFS) was defined as time from initiation of treatment to documented disease progression or death from any cause. progression was defined as the enlargement of the measured sum by 20% or one or more new lesions. This outcome measure was analyzed using Kaplan-Meier method.
Time Frame: From initiation of treatment until the date of first documented progression or date of death from any cause, whichever came first, approximately 13 years and 10 months
Population: Effectiveness analysis set (EAS): all participants included in study with at least 1 information on: date of death, progression, assessment of response to therapy by physician or assessment to either effectiveness or tolerability of therapy by physician. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- mRCC - Temsirolimus: Participants diagnosed with mRCC who received only temsirolimus from January 2008 to December 2021, as per routine clinical practice were observed during this prospective registry study. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with temsirolimus was discontinued or documentation was stopped for any reason.
- mRCC - Sunitinib: Participants diagnosed with mRCC who received sunitinib (some of the participants stopped sunitinib and received axitinib) from January 2008 to December 2021, as per routine clinical practice were observed during this prospective registry study. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with sunitinib was discontinued or documentation was stopped for any reason.
- mRCC - Axitinib: Participants diagnosed with mRCC who received axitinib (some of the participants initially received sunitinib) from January 2008 to December 2021, as per routine clinical practice were observed during this prospective registry study. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with axitinib was discontinued or documentation was stopped for any reason.
- MCL - Temsirolimus: Participants diagnosed with MCL who received only temsirolimus from January 2008 to December 2021, as per routine clinical practice were observed during this prospective registry study. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with temsirolimus was discontinued or documentation was stopped for any reason.
- GIST - Sunitinib: Participants diagnosed with GIST who received only sunitinib from January 2008 to December 2021, as per routine clinical practice were observed during this prospective registry study. Participants in this observational study, were followed up for every 8 to 12 weeks until treatment with sunitinib was discontinued or documentation was stopped for any reason.
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 577 | 651 | 221 | 55 | 24
Months | 11.04 [9.56 to 13.04] | 25.36 [22.18 to 28.22] | 18.37 [14.03 to 24.15] | 15.11 [8.54 to 22.01] | 16.30 [7.29 to 53.22]

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from initiation of treatment to documented disease progression or death from any cause. The presence of a progression i.e. enlargement of the measured sum by 20% or one or more new lesions was confirmed, but (a) No date was documented: the date of last intake of study medication was used as date of progression, otherwise the date of the last visit with a documented "non-progression" was used as date of progression. (b) Dates within a visit and on final documentation were contradictory, the prior date was used. In case a death was documented within survival follow-up, but no progression was documented within regular study, the date of last visit plus 1 day was used as date of progression. In case no progression was documented, participant was censored with the latest available contact date or assessment date within study. In case these rules led to a missing duration or a negative duration, duration was set to "1 day". Kaplan-Meier method was used for analysis.
Time Frame: as for outcome 1
Population: EAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 577 | 651 | 221 | 55 | 24
Months | 3.91 [3.45 to 4.63] | 6.93 [6.24 to 8.25] | 5.75 [4.90 to 6.64] | 3.68 [3.02 to 4.86] | 10.32 [3.58 to 12.94]

3. Primary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR included Complete Remission (CR): complete disappearance of all lesions. Partial Remission (PR): Reduction of the measured total by at least 30%. Minor remission (MR): ≥10% decrease in the sum of longest diameters of target lesions but not a PR (<30%). Stable Disease (SD): neither shrinkage for CR/PR nor increase for progressive disease (PD) taking as reference smallest sum of longest diameters (SLDs) since treatment start. PD: Enlargement of the measured sum by 20% or one or more new lesions. In this outcome measure, number of participants with best overall response were reported.
Time Frame: as for outcome 1
Population: EAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, 'Number Analyzed' signifies those participants who were evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 577 | 651 | 221 | 55 | 24
Participants
  CR | 5 | 40 | 3 | 1 | 0
  PR | 70 | 166 | 39 | 14 | 6
  MR | 0 | 0 | 0 | 3 | 0
  SD | 237 | 221 | 75 | 10 | 11
  PD | 169 | 146 | 58 | 17 | 6
  Response could not be assessed | 88 | 59 | 39 | 10 | 1
  Missing | 8 | 19 | 7 | 0 | 0

4. Primary Outcome: Number of Participants Categorized According to Physician's Global Assessment of Effectiveness
Description: In this outcome measure, number of participants were categorized according to physician's global assessment of effectiveness as very good, good, moderate, insufficient and missing. Categories were determined by investigator's discretion.
Time Frame: as for outcome 1
Population: EAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 505 | 575 | 195 | 48 | 23
Participants
  Very good | 35 | 57 | 6 | 2 | 0
  Good | 176 | 227 | 78 | 20 | 10
  Moderate | 110 | 112 | 43 | 12 | 3
  Insufficient | 159 | 150 | 60 | 12 | 8
  Missing | 25 | 29 | 8 | 2 | 2

5. Primary Outcome: Karnofsky Performance Status (KPS) Scale
Description: Karnofsky performance score was used to quantify participant's general well-being and activities of daily life and participants were classified based on their functional impairment. Karnofsky performance score ranges between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: as for outcome 1
Population: EAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure. This outcome measure was not planned to be analyzed for MCL.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | GIST - Sunitinib
Number analyzed (Participants) | 478 | 547 | 175 | 18
Units on a scale | 71.9 (15.4) | 78.8 (14.1) | 77.9 (13.2) | 77.8 (8.8)

6. Primary Outcome: Number of Participants Classified According to Eastern Cooperative Oncology Group (ECOG) Performance Status for Mantle Cell Lymphoma
Description: ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. In this outcome measure, data for ECOG status (0, 1, 2) and missing was evaluated for MCL as planned.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MCL - Temsirolimus
Number analyzed (Participants) | 48
Participants
  ECOG: 0 | 5
  ECOG: 1 | 24
  ECOG: 2 | 13
  Missing | 6

7. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any undesirable medical event in a participant took a medicinal product. It was not necessarily required that the event is causally related to the treatment or use of the medicinal product. An SAE was any undesirable medical event that occurred in a participant received a medicinal product or dietary supplement (including infant formula) at any dose, and that resulted in death; was life-threatening; required an unforeseen hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial impairment of the ability to perform daily activities); resulted in a congenital malformation/birth defect. TEAEs were events between first dose of study drug and up to last documented follow-up visit that were absent before treatment or that worsened relative to pretreatment state. AEs included serious and all non-serious adverse events.
Time Frame: as for outcome 1
Population: Safety analysis set (SAS) comprised of all prospectively documented participants with histologically proven diagnosis of either mRCC, MCL or GIST and at least 1 documented administration of temsirolimus, sunitinib or axitinib or any non-Pfizer treatment. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study.
Measure: Count of Participants; unit: Participants
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 605 | 702 | 237 | 59 | 26
Participants
  TEAEs | 460 | 585 | 187 | 53 | 20
  SAEs | 269 | 284 | 111 | 26 | 11

8. Primary Outcome: Number of Participants Who Discontinued Treatment Due to Adverse Events
Description: An AE was any undesirable medical event in a participant took a medicinal product. It was not necessarily required that the event is causally related to the treatment or use of the medicinal product. In this outcome measure number of participants who discontinued treatment due to adverse events were reported.
Time Frame: as for outcome 1
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study.
Measure: Count of Participants; unit: Participants
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 605 | 702 | 237 | 59 | 26
Participants | 108 | 142 | 60 | 17 | 5

9. Primary Outcome: Number of Participants Categorized According to Physician's Global Tolerability Assessment
Description: In this outcome measure, number of participants were categorized according to physician's global tolerability assessment as very good, good, moderate, insufficient and missing. Categories were determined by investigator's discretion.
Time Frame: as for outcome 1
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 505 | 576 | 195 | 49 | 24
Participants
  Very good | 93 | 49 | 21 | 5 | 3
  Good | 306 | 370 | 123 | 25 | 16
  Moderate | 68 | 107 | 31 | 13 | 3
  Insufficient | 34 | 40 | 18 | 4 | 0
  Missing | 4 | 10 | 2 | 2 | 2

10. Primary Outcome: Absolute Laboratory Values of Hematology Parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Hematocrit
Time Frame: Week 46 up to Week 55 post study inclusion
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure and 'Number Analyzed' signifies those participants who were evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Percentage of blood cells in blood
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 42 | 115 | 42 | 2 | 8
Percentage of blood cells in blood
  Neutrophils: number analyzed (Participants) | 39 | 102 | 22 | 2 | 8
  Neutrophils | 67.1 (13.2) | 56.0 (14.0) | 64.4 (10.8) | 58.7 (1.0) | 58.7 (13.7)
  Lymphocytes: number analyzed (Participants) | 42 | 107 | 22 | 2 | 8
  Lymphocytes | 18.8 (8.5) | 31.1 (12.0) | 23.7 (9.1) | 22.5 (8.6) | 28.9 (12.6)
  Monocytes: number analyzed (Participants) | 37 | 99 | 22 | 2 | 6
  Monocytes | 8.9 (3.7) | 8.7 (3.3) | 8.4 (2.3) | 14.2 (6.9) | 8.8 (2.9)
  Eosinophils: number analyzed (Participants) | 35 | 88 | 22 | 2 | 5
  Eosinophils | 2.6 (1.9) | 2.9 (2.3) | 3.0 (1.4) | 4.3 (2.8) | 2.1 (2.5)
  Basophils: number analyzed (Participants) | 32 | 88 | 22 | 2 | 5
  Basophils | 0.4 (0.4) | 0.4 (0.3) | 0.5 (0.4) | 0.4 (0.1) | 0.2 (0.1)
  Hematocrit: number analyzed (Participants) | 11 | 115 | 42 | 0 | 0
  Hematocrit | 33.8 (3.5) | 37.0 (5.2) | 42.7 (5.2) |  |

11. Primary Outcome: Absolute Laboratory Values of Hematology Parameters: Hemoglobin A1c (HbA1c)
Time Frame: Week 46 up to Week 55 post study inclusion
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here N=0 signifies that participants were not evaluable at the specified time point for HbA1c in MCL arm.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 3 | 22 | 4 | 0 | 2
Percentage of HbA1c | 7.9 (1.2) | 5.8 (0.8) | 5.9 (0.9) |  | 7.5 (3.2)

12. Primary Outcome: Absolute Laboratory Values of Hematology Parameters: Hemoglobin
Time Frame: Week 46 up to Week 55 post study inclusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 72 | 163 | 45 | 3 | 9
Grams per deciliter | 11.2 (1.6) | 12.2 (2.0) | 14.4 (1.7) | 12.6 (0.8) | 11.9 (1.2)

13. Primary Outcome: Absolute Laboratory Values of Clinical Chemistry Parameters: Calcium, Sodium, Potassium, Phosphate, Magnesium, Cholesterol, Triglycerides and Glucose
Time Frame: Week 46 up to Week 55 post study inclusion
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 63 | 153 | 41 | 2 | 8
Millimoles per liter
  Calcium: number analyzed (Participants) | 63 | 149 | 41 | 2 | 8
  Calcium | 2.3 (0.4) | 2.3 (0.3) | 2.6 (1.1) | 2.4 (0.1) | 2.3 (0.1)
  Sodium: number analyzed (Participants) | 54 | 150 | 35 | 1 | 8
  Sodium | 136.0 (19.1) | 139.1 (3.6) | 138.1 (4.0) | 138.0 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 139.0 (2.7)
  Potassium: number analyzed (Participants) | 56 | 153 | 36 | 2 | 8
  Potassium | 4.3 (0.6) | 4.5 (0.6) | 4.4 (0.6) | 3.6 (0.0) | 4.1 (0.9)
  Phosphate: number analyzed (Participants) | 10 | 60 | 15 | 0 | 3
  Phosphate | 1.4 (0.9) | 1.1 (0.5) | 1.4 (0.9) |  | 0.9 (0.2)
  Magnesium: number analyzed (Participants) | 10 | 39 | 13 | 0 | 1
  Magnesium | 1.2 (0.7) | 0.8 (0.3) | 0.7 (0.1) |  | 0.9 (NA) — Standard deviation was not calculated as only 1 participant was evaluable.
  Cholesterol: number analyzed (Participants) | 18 | 52 | 11 | 0 | 2
  Cholesterol | 6.0 (1.9) | 5.1 (1.3) | 6.6 (1.3) |  | 5.9 (2.1)
  Triglycerides: number analyzed (Participants) | 19 | 56 | 11 | 0 | 2
  Triglycerides | 3.2 (3.4) | 2.4 (1.1) | 3.5 (2.5) |  | 5.2 (3.4)
  Glucose: number analyzed (Participants) | 46 | 99 | 29 | 0 | 4
  Glucose | 54.7 (62.6) | 39.4 (52.4) | 71.4 (78.4) |  | 77.2 (143.2)

14. Primary Outcome: Absolute Laboratory Values of Clinical Chemistry Parameters: Creatinine, Total Bilirubin
Time Frame: Week 46 up to Week 55 post study inclusion
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 54 | 152 | 42 | 2 | 9
Milligrams per deciliter
  Creatinine | 1.4 (0.5) | 1.4 (0.8) | 1.3 (0.5) | 0.7 (0.0) | 1.1 (0.3)
  Total bilirubin: number analyzed (Participants) | 43 | 129 | 33 | 1 | 7
  Total bilirubin | 0.9 (1.7) | 0.7 (1.1) | 0.5 (0.3) | 0.3 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 0.4 (0.1)

15. Primary Outcome: Absolute Laboratory Values of Clinical Chemistry Parameters: Alanine Transaminase (ALT), Aspartate Transaminase (AST), Alkaline Phosphatase (ALP) and Lactate Dehydrogenase (LDH)
Time Frame: Week 46 up to Week 55 post study inclusion
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 52 | 145 | 39 | 1 | 9
Units per liter
  ALT: number analyzed (Participants) | 47 | 145 | 38 | 1 | 9
  ALT | 20.2 (8.3) | 25.9 (17.5) | 34.7 (71.8) | 24.0 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 22.9 (7.5)
  AST: number analyzed (Participants) | 51 | 137 | 35 | 1 | 9
  AST | 23.1 (8.2) | 29.6 (12.8) | 44.3 (84.3) | 28.0 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 24.6 (6.4)
  ALP: number analyzed (Participants) | 48 | 133 | 38 | 1 | 8
  ALP | 95.8 (53.5) | 77.9 (30.6) | 91.8 (43.2) | 130.0 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 79.3 (50.7)
  LDH: number analyzed (Participants) | 52 | 131 | 39 | 1 | 8
  LDH | 224.8 (88.2) | 245.1 (67.2) | 235.8 (126.9) | 256.0 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 227.8 (45.6)

16. Primary Outcome: Absolute Laboratory Values of Clinical Chemistry Parameters: Albumin
Time Frame: Week 46 up to Week 55 post study inclusion
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here N=0 signifies that participants were not evaluable at the specified time point for albumin in MCL arm.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 10 | 76 | 16 | 0 | 1
Grams per liter | 31.1 (17.1) | 33.6 (14.4) | 31.6 (14.8) |  | 42.0 (NA) — Standard deviation was not calculated as only 1 participant was evaluable.

17. Primary Outcome: Absolute Laboratory Values of Clinical Chemistry Parameters: Triiodothyronine (fT3) and Free Thyroxine (fT4)
Time Frame: Week 46 up to Week 55 post study inclusion
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here N=0 signifies that participants were not evaluable at the specified time point for fT3 and fT4 in MCL and GIST arms.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 1 | 46 | 20 | 0 | 0
Picomoles per liter
  fT3: number analyzed (Participants) | 1 | 46 | 19 | 0 | 0
  fT3 | 3.5 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 3.7 (1.0) | 3.8 (1.3) |  |
  fT4: number analyzed (Participants) | 1 | 43 | 20 | 0 | 0
  fT4 | 15.4 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. | 14.8 (4.8) | 13.7 (6.1) |  |

18. Primary Outcome: Absolute Laboratory Values of Clinical Chemistry Parameters: Thyroid Stimulating Hormone (TSH)
Time Frame: Week 46 up to Week 55 post study inclusion
Population: SAS analyzed. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here N=0 signifies that participants were not evaluable at the specified time point for TSH in MCL arm.
Measure: Mean (Standard Deviation); unit: Milliunits per liter
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
Number analyzed (Participants) | 28 | 97 | 27 | 0 | 6
Milliunits per liter | 1.5 (1.4) | 3.5 (3.4) | 3.4 (2.4) |  | 1.6 (1.1)

ADVERSE EVENTS:
Time Frame: Day 1 of study treatment up to last documented follow-up visit, up to 13 years 10 months
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or participant may experienced both a serious and non-serious episode of same event. Participants received another treatment if not benefited from treatment they were receiving at enrollment; participants were not exclusive in few arms. So, sum of participants across arms is not equal to number of participants who started study.
Arm/Group | mRCC - Temsirolimus | mRCC - Sunitinib | mRCC - Axitinib | MCL - Temsirolimus | GIST - Sunitinib
All-Cause Mortality (participants affected / at risk) | 440/605 | 420/702 | 163/237 | 40/59 | 16/26
Serious Adverse Events (participants affected / at risk) | 269/605 | 284/702 | 111/237 | 26/59 | 11/26
Other Adverse Events (participants affected / at risk) | 342/605 | 485/702 | 148/237 | 45/59 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mRCC - Temsirolimus (N=605) | mRCC - Sunitinib (N=702) | mRCC - Axitinib (N=237) | MCL - Temsirolimus (N=59) | GIST - Sunitinib (N=26)
Fatigue (General disorders) | 4 | 6 | 2 | 1 | 0
Disease progression (General disorders) | 66 | 35 | 19 | 4 | 3
General physical health deterioration (General disorders) | 39 | 39 | 16 | 6 | 0
Oedema peripheral (General disorders) | 5 | 2 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 3 | 1 | 1 | 0
Pain (General disorders) | 4 | 7 | 2 | 0 | 0
Pyrexia (General disorders) | 6 | 5 | 1 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 3 | 1 | 0
Condition aggravated (General disorders) | 8 | 2 | 1 | 2 | 0
Chest pain (General disorders) | 2 | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 6 | 2 | 1 | 0 | 0
Impaired healing (General disorders) | 2 | 1 | 1 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0 | 0
Death (General disorders) | 3 | 6 | 7 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 3 | 0 | 0 | 0 | 0
Concomitant disease progression (General disorders) | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 1 | 0
(General disorders) | 0 | 5 | 0 | 0 | 0 — Event was not coded by any medical dictionary and event was captured as Unknown.
Organ failure (General disorders) | 0 | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 8 | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 11 | 13 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 10 | 6 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 0
Ascites (Gastrointestinal disorders) | 7 | 1 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 4 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 5 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oedema mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 11 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 21 | 7 | 4 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 15 | 15 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 11 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 5 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 24 | 19 | 10 | 3 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 3 | 1 | 5 | 0
Infection (Infections and infestations) | 4 | 2 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 3 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 5 | 7 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0 | 1 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Purulence (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Candida pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 3 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 3 | 2 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 2 | 0 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Lipids abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood electrolytes abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 8 | 6 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5 | 3 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 4 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Head titubation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 2 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 5 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2 | 1 | 0 | 1
Paresis (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 2 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 15 | 7 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 27 | 4 | 0 | 3
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 16 | 4 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 6 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 12 | 5 | 4 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 1 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 5 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 2 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cor pulmonale acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bifascicular block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Gastrocardiac syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 8 | 6 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 8 | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0
Renal hypertension (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Vesical fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Postrenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urethral caruncle (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 3 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 2 | 3 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 2 | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic dissection rupture (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Leriche syndrome (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Venous occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 5 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 3 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Arthrectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Nephrectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Leg amputation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mRCC - Temsirolimus (N=605) | mRCC - Sunitinib (N=702) | mRCC - Axitinib (N=237) | MCL - Temsirolimus (N=59) | GIST - Sunitinib (N=26)
Fatigue (General disorders) | 78 | 144 | 39 | 6 | 3
Disease progression (General disorders) | 8 | 14 | 8 | 0 | 0
General physical health deterioration (General disorders) | 16 | 23 | 5 | 5 | 0
Oedema peripheral (General disorders) | 35 | 27 | 1 | 4 | 0
Mucosal inflammation (General disorders) | 27 | 55 | 8 | 4 | 3
Pain (General disorders) | 24 | 13 | 10 | 0 | 0
Pyrexia (General disorders) | 18 | 12 | 3 | 2 | 1
Asthenia (General disorders) | 9 | 11 | 6 | 5 | 0
Condition aggravated (General disorders) | 4 | 2 | 0 | 1 | 0
Oedema (General disorders) | 9 | 13 | 3 | 0 | 0
Chest pain (General disorders) | 5 | 6 | 3 | 1 | 0
Chills (General disorders) | 7 | 8 | 0 | 3 | 1
Feeling cold (General disorders) | 5 | 3 | 1 | 0 | 0
Impaired healing (General disorders) | 2 | 2 | 1 | 0 | 0
Malaise (General disorders) | 3 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 5 | 0 | 0 | 0
Swelling (General disorders) | 4 | 2 | 0 | 1 | 0
Swelling face (General disorders) | 3 | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 2 | 2 | 1 | 0 | 0
Exercise tolerance decreased (General disorders) | 2 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 2 | 2 | 0 | 0 | 0
Generalised oedema (General disorders) | 2 | 0 | 0 | 0 | 0
Chronic fatigue syndrome (General disorders) | 1 | 1 | 0 | 0 | 0
Drug intolerance (General disorders) | 1 | 4 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 3 | 2 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal dryness (General disorders) | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal disorder (General disorders) | 0 | 7 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 2 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 2 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 1 | 0 | 0 | 0
Drug ineffective (General disorders) | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 2 | 0 | 0
Medical device site erosion (General disorders) | 0 | 1 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 1 | 0 | 0 | 0
No adverse event (General disorders) | 0 | 0 | 2 | 0 | 0
Gait inability (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal pain (General disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 47 | 89 | 19 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 29 | 149 | 64 | 12 | 6
Vomiting (Gastrointestinal disorders) | 22 | 37 | 10 | 5 | 2
Stomatitis (Gastrointestinal disorders) | 26 | 68 | 9 | 3 | 3
Ascites (Gastrointestinal disorders) | 10 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 14 | 19 | 8 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 10 | 9 | 4 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 14 | 6 | 2 | 1
Aphthous ulcer (Gastrointestinal disorders) | 7 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 5 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 3 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 6 | 4 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 41 | 3 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 5 | 2 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 10 | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oedema mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Tongue exfoliation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Tongue discomfort (Gastrointestinal disorders) | 0 | 7 | 2 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tongue blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tongue erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 | 40 | 11 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 29 | 10 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 26 | 3 | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 19 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 83 | 61 | 9 | 13 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 73 | 2 | 24 | 5
Leukopenia (Blood and lymphatic system disorders) | 20 | 68 | 1 | 12 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 8 | 0 | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2 | 3 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Erythropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 6 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 4 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 14 | 7 | 3 | 2 | 0
Urinary tract infection (Infections and infestations) | 13 | 8 | 6 | 3 | 1
Infection (Infections and infestations) | 10 | 6 | 2 | 3 | 0
Nasopharyngitis (Infections and infestations) | 13 | 15 | 2 | 3 | 1
Erysipelas (Infections and infestations) | 4 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 6 | 1 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 5 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 5 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Candida infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 3 | 3 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 2 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 1 | 1 | 1 | 0
Febrile infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Pustule (Infections and infestations) | 2 | 1 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Acne pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Fungal foot infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection susceptibility increased (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Superinfection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anal fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 44 | 21 | 13 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 19 | 6 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 12 | 9 | 0 | 2 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 | 85 | 17 | 1 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 13 | 2 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 8 | 3 | 2 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 8 | 2 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 6 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9 | 4 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 6 | 2 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 4 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 5 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Epidermolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 13 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 26 | 28 | 7 | 1 | 0
Haemoglobin decreased (Investigations) | 29 | 9 | 0 | 2 | 0
Weight decreased (Investigations) | 11 | 33 | 21 | 2 | 1
Blood glucose increased (Investigations) | 11 | 3 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 10 | 11 | 5 | 2 | 0
Blood cholesterol increased (Investigations) | 7 | 1 | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 6 | 4 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 5 | 0 | 2 | 0 | 0
Platelet count decreased (Investigations) | 5 | 2 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 3 | 3 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 3 | 26 | 5 | 0 | 0
Body temperature increased (Investigations) | 3 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 4 | 2 | 0 | 0
Platelet count increased (Investigations) | 3 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 3 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 7 | 2 | 0 | 0
Blood albumin decreased (Investigations) | 2 | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 2 | 19 | 6 | 1 | 0
Blood sodium decreased (Investigations) | 2 | 0 | 1 | 0 | 0
Blood triglycerides abnormal (Investigations) | 2 | 1 | 0 | 0 | 0
Haemoglobin (Investigations) | 2 | 0 | 0 | 0 | 0
Lipids increased (Investigations) | 2 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 2 | 3 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 2 | 2 | 0 | 0 | 0
Amylase abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 7 | 4 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 3 | 0 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood cholesterol abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 1 | 3 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine (Investigations) | 1 | 1 | 0 | 0 | 0
Blood immunoglobulin M decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 2 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 2 | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 1 | 1 | 0 | 0 | 0
Computerised tomogram thorax abnormal (Investigations) | 1 | 1 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 1 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 1 | 0 | 0 | 0
Quality of life decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 1 | 0 | 0 | 0
White blood cell count (Investigations) | 1 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 3 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 3 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 3 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 3 | 3 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Blood glucose (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood uric acid abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Thyroxine free increased (Investigations) | 0 | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 26 | 68 | 21 | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3 | 2 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 2 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 5 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 7 | 2 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 5 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 7 | 2 | 0 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 17 | 26 | 8 | 0 | 1
Taste disorder (Nervous system disorders) | 14 | 74 | 3 | 1 | 3
Headache (Nervous system disorders) | 12 | 19 | 7 | 1 | 1
Paraesthesia (Nervous system disorders) | 6 | 6 | 3 | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 12 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 3 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 2 | 3 | 2 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 3 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 1 | 26 | 2 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 2 | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 3 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 4 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrospinal fluid retention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Clumsiness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6 | 4 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 12 | 3 | 0 | 0
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 3 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 22 | 13 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 21 | 8 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 28 | 8 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 9 | 5 | 3 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 9 | 3 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 8 | 2 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bone loss (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 2 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 1 | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Cardiac flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiotoxicity (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Rhythm idioventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 6 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 4 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 63 | 14 | 0 | 1
Lymphoedema (Vascular disorders) | 5 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 3 | 5 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 6 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 4 | 2 | 0 | 0
Thrombosis (Vascular disorders) | 3 | 2 | 0 | 0 | 0
Hot flush (Vascular disorders) | 2 | 2 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Fibromuscular dysplasia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Jugular vein distension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Subclavian artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin pressure mark (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Off label use (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 6 | 4 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 3 | 12 | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 2 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Tobacco abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Transient psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0
Claustrophobia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Sleep attacks (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 4 | 9 | 0 | 0 | 0
Visual impairment (Eye disorders) | 3 | 2 | 1 | 0 | 0
Eye irritation (Eye disorders) | 2 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 4 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 2 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 2 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 2 | 0 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye paraesthesia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 5 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion removal (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Red blood cell transfusion (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Stent removal (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 3 | 0 | 0 | 0
Ankle operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Hyperthermia therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Jaw operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 7 | 1 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 30 | 16 | 0 | 1
Thyroid disorder (Endocrine disorders) | 1 | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 2 | 3 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Genital tract inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Contrast media reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Corneal graft rejection (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Product supply issue (Product Issues) | 0 | 0 | 1 | 0 | 0
Bedridden (Social circumstances) | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT00700258/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT00700258/SAP_001.pdf